CLINICAL TRIAL: NCT07006701
Title: A Population-based Cohort of Osteoarthritis: the Tsinghua University Tiantongyuan Community Osteoarthritis Study
Status: Not yet recruiting | Type: Observational
Sponsor: Beijing Tsinghua Chang Gung Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 25025-4-01
Record Dates: First submitted 2025-05-20; First posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The purpose of this study is to examine the natural history and risk factors of osteoarthritis (OA) and to explore the relationship between metabolic factors and OA progression.

DETAILED DESCRIPTION:
1. To investigate the natural history of osteoarthritis (OA) in a large-sample cohort.
2. To identify OA phenotypes and their relationship with clinical symptoms and functional impairment.
3. To analyze metabolic factors (e.g., obesity, diabetes, and hypertension) as risk factors for OA onset and progression.
4. To evaluate the association between radiographic changes and OA symptoms.
5. To develop predictive models for OA progression and identify high-risk individuals for early intervention.

Design: This is a prospective cohort study. Participants: The study will recruit approximately 4,000 individuals aged 50 years and above. Participants will undergo baseline assessments, including demographic data collection, medical history, dietary evaluation, physical examination, blood sample collection, and radiographic imaging. Annual follow-ups will be conducted over 10 years to monitor OA progression and related risk factors.

ELIGIBILITY:
Inclusion Criteria:

* Aged 50 years and above
* Long-term resident of the study area
* Willing to participate and provide informed consent

Exclusion Criteria:

* Hearing, speech, or mental impairments preventing effective communication
* Unable to complete scheduled follow-up visits
* Pregnant or planning pregnancy during the study period
* Any other condition deemed unsuitable for participation by the researchers

Min Age: 50 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This study will include adults aged 50 years and above to investigate osteoarthritis risk factors and progression in a general population-based cohort.
Sampling Method: Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2025-06-03 (Estimated); Primary Completion 2034-12-31 (Estimated); Study Completion 2034-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Osteoarthritis | Annually for 10 years
  The occurrence of clinically diagnosed osteoarthritis based on imaging and clinical symptoms during the follow-up period.

SECONDARY OUTCOMES:
Change in Joint Pain Severity (WOMAC Pain Subscale) | Annually for 10 years
  Evaluated using the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) pain subscale (range: 0-20). Higher scores indicate worse pain.
Change in Physical Function (WOMAC Subscale) | Annually for 10 years
  Assessed using the WOMAC physical function subscale (range: 0-68). Higher scores indicate worse physical function.
Change in Physical Function (SF-36 Physical Function Domain) | Annually for 10 years
  Assessed using the SF-36 physical function domain (range: 0-100). Higher scores indicate better physical function.
Timed Up and Go Test (TUGT) | Annually for 10 years
  Measured in seconds; a shorter time indicates better mobility.
Five Times Sit-to-Stand Test (5TSTS) | Annually for 10 years
  Measured in seconds; a shorter time indicates better lower limb strength and function.
Radiographic Progression of Osteoarthritis | Annually for 10 years
  Measured by changes in Kellgren-Lawrence (K-L) grade in bilateral knee X-rays over time.
Changes in Body Mass Index (BMI) | Annually for 10 years
  Measured in kg/m². Analyzed for correlation with radiographic progression of osteoarthritis using the Kellgren-Lawrence grading system.
Changes in Blood Pressure | Annually for 10 years
  Measured in mmHg using an automated sphygmomanometer to record systolic and diastolic blood pressure.
Changes in Fasting Glucose | Annually for 10 years
  Measured in mg/dL using venous blood samples collected after an overnight fast.
Changes in Total Cholesterol (TC) | Annually for 10 years
  Measured in mmol/L or mg/dL using fasting venous blood samples.
Changes in Low-Density Lipoprotein Cholesterol (LDL-C) | Annually for 10 years
  Measured in mmol/L or mg/dL using fasting venous blood samples.
Changes in High-Density Lipoprotein Cholesterol (HDL-C) | Annually for 10 years
  Measured in mmol/L or mg/dL using fasting venous blood samples.
Changes in Triglycerides (TG) | Annually for 10 years
  Measured in mmol/L or mg/dL using fasting venous blood samples.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tsinghua Chang Gung Hospital, Beijing, Beijing Municipality, China